CLINICAL TRIAL: NCT00283439
Title: An Open Label Dose and Schedule Finding Trial to Evaluate the Safety and Efficacy of AMG 531 for Treatment of Severe Thrombocytopenia Due to Multi-Cycle Chemotherapy in Adult Subjects With Lymphoma.
Brief Title: A Dose and Schedule Finding Trial With AMG 531 for Chemotherapy Induced Thrombocytopenia (CIT) in Adults With Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20050144
Record Dates: First submitted 2006-01-26; First posted 2006-01-30 (Estimated); Results first posted 2010-09-13 (Estimated); Last update posted 2011-06-20 (Estimated); Status verified 2011-06

CONDITIONS: Chemotherapy-Induced Thrombocytopenia; Hodgkin's Lymphoma; Non-Hodgkin's Lymphoma; Cancer; Oncology; Thrombocytopenia
Keywords: NHL; chemotherapy induced thrombocytopenia; CIT; ICE; RICE; Hodgkin's Lymphoma; Non-Hodgkin's Lymphoma; CHOP; ESHAP; DHAP; R-CHOP; R-ESHAP; R-DHAP
MeSH Terms: conditions — Hodgkin Disease; Lymphoma, Non-Hodgkin; Neoplasms; Thrombocytopenia | interventions — romiplostim

ARMS (1):
- Single Arm: AMG 531 Dose-Escalating Cohort Study (Experimental)
  Interventions: Biological: AMG 531

INTERVENTIONS:
Biological: AMG 531 — Planned Cohorts:
  1. 100 mcg,
  2. 300 mcg,
  3. 700 mcg,
  4. 1000 mcg;
     Optional Cohorts:
  5. cohort expansion,
  6. schedule change,
  7. new dose

SUMMARY:
The purpose of this study is to identify a well-tolerated, effective dose and schedule of AMG 531 for the treatment of Chemotherapy Induced Thrombocytopenia (CIT) in subjects with lymphoma receiving multi-cycle chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed Hodgkin's lymphoma or Non-Hodgkin's lymphoma receiving Q14, Q21, or Q28 day CHOP, ICE, ESHAP, or DHAP chemotherapy; with or without Rituximab
* Has adequate bone marrow function; platelet count > 100 x 10^9/L on the day of initiation of the on study chemotherapy of the next treatment cycle and absolute neutrophil count, ANC > or = 1 x 10^9/L, and hemoglobin > or = 9.5 g/dL
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Has adequate liver function
* must be able to receive the same chemotherapy regimen during the first treatment cycle as was received during the prior qualifying cycle
* must experience Common Terminology Criteria (CTC) grade 3 or 4 thrombocytopenia (platelet count < 50 x 10^9/L) as a result of the chemotherapy administered in the cycle immediately preceding study entry
* has serum creatinine concentration < or = 2 mg/dl

Exclusion Criteria:

* More that 1 prior relapse chemotherapy regimen
* Sepsis, disseminated coagulation or any other condition that may exacerbate thrombocytopenia
* Significant bleeding (CTC grade 3 or 4)
* History of thromboembolic disease
* Subjects who are identified by clinical history and/or serological testing to have either acute or chronic hepatitis B or C infection or to be HIV positive
* Use of any nitrosourea or mitomycin-C
* Has received any thrombocytopenic growth factor
* Has received a marrow or peripheral blood stem cell infusion
* Known hypersensitivity to any recombinant E. coli-derived product

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2005-10; Primary Completion 2008-05 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com
- See also: Notice regarding posted summaries of trial results — http://download.veritasmedicine.com/REGFILES/amgen/Amgen_results_disclaimer.pdf
- See also: FDA-approved Drug Labeling — http://www.nplate.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 15 March 2006 through 28 April 2008
Groups:
- Romiplostim 100 µg: Romiplostim 100 µg administered by subcutaneous injection on the first day after chemotherapy
- Romiplostim 300 µg: Romiplostim 300 µg administered by subcutaneous injection on the first day after chemotherapy
- Romiplostim 700 µg: Romiplostim 700 µg administered by subcutaneous injection on the first day after chemotherapy
- Romiplostim 1000 µg: Romiplostim 1000 µg administered by subcutaneous injection on the first day after chemotherapy
Period: Overall Study
Arm/Group | Romiplostim 100 µg | Romiplostim 300 µg | Romiplostim 700 µg | Romiplostim 1000 µg
Started | 8 | 11 | 11 | 9
Completed | 0 | 0 | 0 | 0
Not Completed | 8 | 11 | 11 | 9
Not completed — Adverse Event | 0 | 0 | 0 | 1
Not completed — Death | 0 | 0 | 1 | 0
Not completed — Disease progression | 0 | 1 | 0 | 0
Not completed — Requirement for alternative therapy | 1 | 2 | 5 | 2
Not completed — Stem cell transplant | 6 | 6 | 4 | 3
Not completed — Treatment discontinued | 0 | 2 | 1 | 3
Not completed — Other | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Romiplostim 100 µg | Romiplostim 300 µg | Romiplostim 700 µg | Romiplostim 1000 µg | Total
Number analyzed (Participants) | 8 | 11 | 11 | 9 | 39
Age Continuous [Mean (Standard Deviation); unit: Year] | 61.3 (6.2) | 58.1 (9.5) | 54.0 (16.3) | 59.9 (10.6) | 58.0 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 4 | 5 | 15
  Male | 5 | 8 | 7 | 4 | 24
Race/Ethnicity, Customized [Number; unit: Participant]
  White or Caucasian | 6 | 10 | 10 | 8 | 34
  Black or African American | 0 | 0 | 1 | 1 | 2
  Hispanic or Latino | 2 | 1 | 0 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Change in Platelet Nadir
Description: Change in platelet nadir from the previous qualifying cycle to the first treatment cycle.
Time Frame: 32 weeks
Population: Efficacy Analysis Set, composed of all enrolled participants who received at least one dose of romiplostim, completed the first treatment cycle, and were not replaced per the protocol.
Measure: Mean (Standard Error); unit: 10^9/L
Arm/Group | Romiplostim 100 µg | Romiplostim 300 µg | Romiplostim 700 µg | Romiplostim 1000 µg
Number analyzed (Participants) | 8 | 11 | 10 | 9
10^9/L | 17.1 (8.3) | 11.2 (6.1) | 5.1 (6.1) | -5.2 (7.8)
Statistical Analysis 1: Comparison: Romiplostim 100 µg vs Romiplostim 1000 µg; Test type: Superiority or Other; p = 0.9654, Satterhwaite t-test — One-sided test
Statistical Analysis 2: Comparison: Romiplostim 100 µg vs Romiplostim 700 µg; Test type: Superiority or Other; p = 0.8690, Satterhwaite t-test — One-sided test
Statistical Analysis 3: Comparison: Romiplostim 100 µg vs Romiplostim 300 µg; Test type: Superiority or Other; p = 0.7133, Satterhwaite t-test — One-sided test

2. Secondary Outcome: Percentage of Subjects Experiencing Grade 3 or 4 Thrombocytopenia
Description: Percentage of subjects experiencing grade 3 and/or 4 thrombocytopenia (<50 x 10^9/L, and <25 x 10^9/L)
Time Frame: 32 weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Romiplostim 100 µg | Romiplostim 300 µg | Romiplostim 700 µg | Romiplostim 1000 µg
Number analyzed (Participants) | 8 | 11 | 10 | 9
Percentage of participants | 62.5 | 81.8 | 80.0 | 88.9
Statistical Analysis 1: Comparison: Romiplostim 100 µg vs Romiplostim 1000 µg; Test type: Superiority or Other; p = 0.294, Fisher Exact
Statistical Analysis 2: Comparison: Romiplostim 100 µg vs Romiplostim 700 µg; Test type: Superiority or Other; p = 0.608, Fisher Exact
Statistical Analysis 3: Comparison: Romiplostim 100 µg vs Romiplostim 300 µg; Test type: Superiority or Other; p = 0.603, Fisher Exact

3. Secondary Outcome: Duration of Grade 3 or 4 Thrombocytopenia
Description: Duration of grade 3 and/or 4 thrombocytopenia (<50 x 10^9/L and <25 x 10^9/L, respectively)
Time Frame: 32 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Day
Arm/Group | Romiplostim 100 µg | Romiplostim 300 µg | Romiplostim 700 µg | Romiplostim 1000 µg
Number analyzed (Participants) | 8 | 11 | 10 | 9
Day | 3.9 (1.3) | 3.6 (0.9) | 6.0 (1.5) | 8.3 (2.1)
Statistical Analysis 1: Comparison: Romiplostim 100 µg vs Romiplostim 1000 µg; Test type: Superiority or Other; p = 0.091, Satterhwaite t-test
Statistical Analysis 2: Comparison: Romiplostim 100 µg vs Romiplostim 700 µg; Test type: Superiority or Other; p = 0.300, Satterhwaite t-test
Statistical Analysis 3: Comparison: Romiplostim 100 µg vs Romiplostim 300 µg; Test type: Superiority or Other; p = 0.881, Satterhwaite t-test

4. Secondary Outcome: Percentage of Subjects That Received Platelet Transfusions
Description: Percentage of subjects that received platelet transfusions during the first romiplostim treatment cycle
Time Frame: 32 weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Romiplostim 100 µg | Romiplostim 300 µg | Romiplostim 700 µg | Romiplostim 1000 µg
Number analyzed (Participants) | 8 | 11 | 10 | 9
Percentage of participants | 12.5 | 0.0 | 30.0 | 33.3
Statistical Analysis 1: Comparison: Romiplostim 100 µg vs Romiplostim 1000 µg; Test type: Superiority or Other; p = 0.576, Fisher Exact
Statistical Analysis 2: Comparison: Romiplostim 100 µg vs Romiplostim 700 µg; Test type: Superiority or Other; p = 0.588, Fisher Exact
Statistical Analysis 3: Comparison: Romiplostim 100 µg vs Romiplostim 300 µg; Test type: Superiority or Other; p = 0.421, Fisher Exact

ADVERSE EVENTS:
Time Frame: From the first administration of investigation product through 30 days after the last dose of investigational product or end of the study (including the follow-up period), whichever is longer.
Description: The table of Other Adverse Events summarizes the most frequent non-serious occurrences of adverse events.
Arm/Group | Romiplostim 100 µg | Romiplostim 300 µg | Romiplostim 700 µg | Romiplostim 1000 µg
Serious Adverse Events (participants affected / at risk) | 0/8 | 1/11 | 3/11 | 3/9
Other Adverse Events (participants affected / at risk) | 6/8 | 9/11 | 7/11 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Romiplostim 100 µg (N=8) | Romiplostim 300 µg (N=11) | Romiplostim 700 µg (N=11) | Romiplostim 1000 µg (N=9)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 1
Device related infection (Infections and infestations) | 0 | 1 | 0 | 0
Staphylococcal infection (Infections and infestations) | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Convulsion (Nervous system disorders) | 0 | 0 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Romiplostim 100 µg (N=8) | Romiplostim 300 µg (N=11) | Romiplostim 700 µg (N=11) | Romiplostim 1000 µg (N=9)
Anaemia (Blood and lymphatic system disorders) | 1 | 3 | 0 | 3
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2
Diastolic dysfunction (Cardiac disorders) | 0 | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Vision blurred (Eye disorders) | 0 | 1 | 1 | 0
Visual disturbance (Eye disorders) | 0 | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 2 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Hyperchlorhydria (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 5 | 1 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Rectal fissure (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Asthenia (General disorders) | 0 | 1 | 0 | 0
Catheter site pain (General disorders) | 0 | 0 | 1 | 1
Catheter site related reaction (General disorders) | 0 | 0 | 0 | 1
Fatigue (General disorders) | 1 | 2 | 1 | 4
Influenza like illness (General disorders) | 0 | 0 | 0 | 1
Oedema peripheral (General disorders) | 1 | 0 | 0 | 3
Pain (General disorders) | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 2
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 1 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 1 | 0 | 1
Rhinitis (Infections and infestations) | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Back injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 2
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 1
Headache (Nervous system disorders) | 1 | 1 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 0 | 0
Tremor (Nervous system disorders) | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 2 | 0 | 0 | 0
Chromaturia (Renal and urinary disorders) | 0 | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 1 | 0 | 0 | 2
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
Nocturia (Renal and urinary disorders) | 0 | 1 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
Urine flow decreased (Renal and urinary disorders) | 0 | 1 | 0 | 0
Penile oedema (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Increased tendency to bruise (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Haematopoietic stem cell mobilisation (Surgical and medical procedures) | 0 | 0 | 1 | 0
Flushing (Vascular disorders) | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multi-center studies, the investigator agrees not to publish any results before the first multi-center publication.